CLINICAL TRIAL: NCT05783219
Title: Lidocaine Patches Prior to Percutaneous Nerve Evaluation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Stacy Lenger MD, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22.0973
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Overactive Bladder; Urge Incontinence; Fecal Incontinence
Keywords: lidocaine
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: This is a single-center, double-blinded, placebo-controlled, randomized trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized with a stratified block randomization scheme (with a random block size of 4, 6, and 8 participants). Randomization sequence will be generated by statistician collaborator
  A patch (intervention or control) will be removed by a medical assistant prior to provider entering the room in order to secure blinding. 1% lidocaine 10cc will be injected into the sacral procedure site for adequate pain relief. PNE procedure will then be performed. If inadequate analgesia is reported by the Patient during the procedure, additional injectable lidocaine will be administered in 5 cc increments, not to exceed 4.5 mg/kg of injectable lidocaine. The volume of injectable lidocaine used will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- topical lidocaine patch (Experimental): 4% lidocaine patch placed over the sacrum 30 minutes prior to PNE procedure
  Interventions: Drug: Lidocaine patch
- Placebo (Placebo Comparator): Adhesive patch placed over the sacrum 30 minutes prior to PNE procedure
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine patch — 4% lidocaine patch placed over the sacrum 30 minutes prior to PNE procedure
  Arms: topical lidocaine patch
Other: Placebo — Adhesive patch placed over the sacrum 30 minutes prior to PNE procedure
  Arms: Placebo

SUMMARY:
The study will be a double-blind randomized control trial comparing 4% lidocaine patch placed over the sacrum 3 minutes prior to a percutaneous nerve evaluation (PNE) procedure to a placebo patch in patients already scheduled to undergo a medically indicated percutaneous nerve evaluation (PNE). VAS pain score, The volume of injectable lidocaine used, Patient Satisfaction Score, rate of successful PNE (defined as successful placement of wire in the S3 spinal foramen), and the amplitude of perineal stimulation on a Likert scale will be collected immediately after the procedure. Patients will follow up in 1 week - as is standard of care with the PNE procedure. Adverse events such as pain or change in sensation will be recorded. Number of voids and incontinence episodes per day after the PNE procedure will be recorded. Overall satisfaction score will be recorded at that time. Rate of progression to Sacral nerve stimulator implantation will be collected.

The investigators hypothesize that patients in the lidocaine patch group will experience significantly less pain at the time of PNE as measured by a lower change in VAS pain score when compared with the control group.

DETAILED DESCRIPTION:
The study design will be a double-blind randomized control trial comparing 4% lidocaine patch placed over the sacrum 30 minutes prior to the procedure to placebo patch. Intervention and control patches will be in envelopes labeled with study number and located within the procedure area. A patch from the envelope corresponding to the patient will be placed by a medical assistant or co-investigator who is not associated with the PNE placement procedure 30 minutes prior to the procedure start. Number of voids and incontinence episodes per day prior to the PNE procedure will be recorded. A patch (intervention or control) will be removed by a medical assistant prior to provider entering the room in order to secure blinding. 1% lidocaine 10cc will be injected into the sacral procedure site for adequate pain relief. PNE procedure will then be performed. If inadequate analgesia is reported by the Patient during the procedure, additional injectable lidocaine will be administered in 5 cc increments, not to exceed 4.5 mg/kg of injectable lidocaine. The volume of injectable lidocaine used will be recorded. VAS pain scores prior to and immediately after procedure will be recorded. Patient Satisfaction Score, rate of successful PNE, rate of progression to SNS implantation, and amplitude of perineal stimulation of a Likert scale will be collected immediately after the procedure.

Patients will follow up in 1 week - as is standard of care with the PNE procedure. Adverse events such as pain or change in sensation will be recorded. Number of voids and incontinence episodes per day after the PNE procedure will be recorded. The overall satisfaction score will be recorded at that time.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients undergoing sacral neuromodulation to manage their OAB with sacral neuromodulation trial with percutaneous nerve evaluation (PNE) without fluoroscopy.
2. No contraindication to the use of lidocaine patch
3. Age >18 years old

Exclusion Criteria:

1. Patients who are not candidates for SNM therapy
2. Patients with contraindications to SNM including pregnancy
3. Allergy to lidocaine or adhesives
4. Chronic pain as an indication for the PNE procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ULP Female Pelvic Medicine and Reconstructive Surgery - Springs Medical Center Suite 190, Louisville, Kentucky
  - ULP Female Pelvic Medicine and Reconstructive Surgery - Urogynecology Associates office, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Goldman HB, Lloyd JC, Noblett KL, Carey MP, Castano Botero JC, Gajewski JB, Lehur PA, Hassouna MM, Matzel KE, Paquette IM, de Wachter S, Ehlert MJ, Chartier-Kastler E, Siegel SW. International Continence Society best practice statement for use of sacral neuromodulation. Neurourol Urodyn. 2018 Jun;37(5):1823-1848. doi: 10.1002/nau.23515. Epub 2018 Apr 11. PMID 29641846
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Schlenk EA, Erlen JA, Dunbar-Jacob J, McDowell J, Engberg S, Sereika SM, Rohay JM, Bernier MJ. Health-related quality of life in chronic disorders: a comparison across studies using the MOS SF-36. Qual Life Res. 1998 Jan;7(1):57-65. doi: 10.1023/a:1008836922089. PMID 9481151
- [Background] Gormley EA, Lightner DJ, Burgio KL, Chai TC, Clemens JQ, Culkin DJ, Das AK, Foster HE Jr, Scarpero HM, Tessier CD, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline. J Urol. 2012 Dec;188(6 Suppl):2455-63. doi: 10.1016/j.juro.2012.09.079. Epub 2012 Oct 24. PMID 23098785
- [Background] Gupta P, Ehlert MJ, Sirls LT, Peters KM. Percutaneous tibial nerve stimulation and sacral neuromodulation: an update. Curr Urol Rep. 2015 Feb;16(2):4. doi: 10.1007/s11934-014-0479-1. PMID 25630918
- [Background] Siegel S, Noblett K, Mangel J, Bennett J, Griebling TL, Sutherland SE, Bird ET, Comiter C, Culkin D, Zylstra S, Kan F, Berg KC. Five-Year Followup Results of a Prospective, Multicenter Study of Patients with Overactive Bladder Treated with Sacral Neuromodulation. J Urol. 2018 Jan;199(1):229-236. doi: 10.1016/j.juro.2017.07.010. Epub 2017 Jul 11. PMID 28709886
- [Background] Gammaitoni AR, Alvarez NA, Galer BS. Safety and tolerability of the lidocaine patch 5%, a targeted peripheral analgesic: a review of the literature. J Clin Pharmacol. 2003 Feb;43(2):111-7. doi: 10.1177/0091270002239817. PMID 12616661
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Derived] Rothenberger RW, Henry T, Carbone L, Gaskins JT, Gupta A, Francis S, Lenger SM. Supplemental Lidocaine Patches Prior to Percutaneous Nerve Evaluation, a Randomized Trial. Urogynecology (Phila). 2025 Apr 1;31(4):377-383. doi: 10.1097/SPV.0000000000001624. Epub 2025 Feb 25. PMID 40013530

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Lidocaine Patch: 4% lidocaine patch placed over the sacrum 30 minutes prior to PNE procedure
  Lidocaine patch: 4% lidocaine patch placed over the sacrum 30 minutes prior to PNE procedure
  20 participants received the 4% lidocaine patch
- Placebo: Adhesive patch placed over the sacrum 30 minutes prior to PNE procedure
  Placebo: Adhesive patch placed over the sacrum 30 minutes prior to PNE procedure
  19 participants received the 4% lidocaine patch
Period: Overall Study
Arm/Group | Topical Lidocaine Patch | Placebo
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Lidocaine Patch | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 10 | 27
  >=65 years | 3 | 9 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (16) | 57 (10) | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 16 | 18 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Score
Description: Visual Analog Scale pain score (indicating the difference between pre and post-procedural pain scores). The scores in question were 100 mm visual analog scale pain scores. This scale ranges from 0-100mm. Higher 100mm Visual Analog Scale pain scores indicate worsening pain.
Time Frame: collected before and immediately after the PNE procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Topical Lidocaine Patch | Placebo
Number analyzed (Participants) | 20 | 19
mm | 45 (17) | 61 (21)

2. Secondary Outcome: Overall Satisfaction
Description: Satisfaction score collected after PNE procedure. This was accomplished by a Likert scale ranging from "not satisfied" to "somewhat satisfied" to "moderately satisfied" to "quite a bit satisfied". with increasing answers indicating increased satisfaction with the Percutaneous nerve evaluation procedural experience.
Time Frame: immediately after PNE procedure
Measure: Number; unit: Participants
Arm/Group | Topical Lidocaine Patch | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Not Satisfied | 0 | 0
  Somewhat Satisfied | 2 | 3
  Moderately Satisfied | 4 | 7
  Quite A Bit Satisfied | 14 | 9

3. Secondary Outcome: Volume of Injectable Lidocaine Used
Description: The volume in milliliters of injectable lidocaine used for analgesia with the PNE procedure
Time Frame: collected after the PNE procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Topical Lidocaine Patch | Placebo
Number analyzed (Participants) | 20 | 19
mL | 12.7 (4.7) | 13.4 (5.8)

4. Secondary Outcome: Amplitude of Perineal Sensation.
Description: Amplitude of perineal sensation during the PNE procedure. This was accomplished with a 100mm Visual analog scale score. This scale had 0mm indicating no sensation through 100mm indicating the most sensation one has ever felt. This was assessed during percutaneous nerve evaluation stimulation. The aim of the percutaneous nerve evaluation procedure is to achieve high sensation in the region of interest during stimulation - a proxy for appropriate lead placement. Thus, high values on this 100mm Visual analog scale indicate a better outcome.
Time Frame: collected immediately after the PNE procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Topical Lidocaine Patch | Placebo
Number analyzed (Participants) | 20 | 19
mm | 48 (27) | 41 (24)

5. Secondary Outcome: Rate of Successful PNE
Description: Rate of successful stimulation and lead placement with the PNE procedure
Time Frame: collected immediately after the PNE procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Lidocaine Patch | Placebo
Number analyzed (Participants) | 20 | 19
Participants | 20 | 19

6. Secondary Outcome: Rate of Progression to Permanent SNS Implantation
Description: The rate of successful reduction in urinary or fecal incontinence symptoms meriting placement of permanent sacral nerve stimulator
Time Frame: to be assessed 6 months after the PNE procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Lidocaine Patch | Placebo
Number analyzed (Participants) | 20 | 19
Participants | 14 | 13

ADVERSE EVENTS:
Time Frame: 6 months post-procedure
Description: For this study, the following standard adverse event (AE) definitions are used:
  * Adverse event: Any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medical treatment or procedure, regardless of relatedness to the treatment
  * Serious Adverse Event (SAE): Any AE related to the study drug that results in: death, life-threatening, event requiring inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability
Arm/Group | Topical Lidocaine Patch | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT05783219/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT05783219/ICF_001.pdf